CLINICAL TRIAL: NCT05042531
Title: Clinical Research for Azacitidine Combined With Low-dose Dasatinib in Maintenance Therapy of Acute Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Collaborators: Beijing Health Alliance Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Bei Liu, Chief Physician, Clinical Associate Professor，Deputy Director of Hematology Department, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZALDDASA3; ChiCTR2100042418 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML,Maintenance Therapy,Azacitidine,Dasatinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Dasatinib

STUDY DESIGN:
Intervention Model Description: The patients were randomly divided into two groups among intermediate and high-risk AML, namely azacitidine group, azacitidine combined with low-dose dasatinib group, with overall survival and disease-free survival as the main research endpoints , taking mortality and recurrence rates as secondary research endpoints, assessing the incidence of adverse events, and studying its related mechanisms.
Who Masked: Investigator
Masking Description: According to the random number table
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients with intermediate and high risk AML were negative for minimal residual disease after intensive induction and consolidation chemotherapy,the patients were randomly divided into two groups, and one group was given azacitidine(75mg/m2, per day on day 1-7]. Dasatinib 100 mg p.o. qd was administered on days 1-28 of each consolidation cycle.
  Interventions: Drug: Azacitidine; Drug: Dasatinib
- control group (Active Comparator): Patients with intermediate and high risk AML were negative for minimal residual disease after intensive induction and consolidation chemotherapy,the patients were randomly divided into two groups, and the other group was given azacitidine(75mg/m2, per day on day 1-7)on days 1-28 of each consolidation cycle.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine, 75mg/m2,d1-7;Treatment cycles every 28 days
Drug: Dasatinib — dasatinib,20mg,po,qd,treatment cycles every 28 days
  Arms: experimental group

SUMMARY:
This project is a prospective, single-center study to evaluate the efficacy, safety and related mechanisms of azacitidine combined with low-dose dasatinib in maintenance therapy in patients with intermediate and high-risk acute myeloid leukemia(AML). The patients were randomly divided into azacitidine group and azacitidine combined with low-dose dasatinib group. The overall survival and disease-free survival were taken as the main end points, and the mortality and recurrence rate were taken as the secondary end points, meanwhile, the incidence of adverse events were evaluated. At the same time, the mRNA expressions of DNA methyltransferase (DNMT1, DNMT3a, DNMT3b), tumor suppressor genes (TP53, P15, P16, P21, CDH1, DOK6, SHP1, PTPN11) and differentiation genes (pu.1, C/EBP α, C/EBP β) were detected. Pyrophosphate sequencing was used to detect the methylation level of the promoter region of these tumor suppressor genes. Western Blot was used to detect apoptosis proteins (caspase3, caspase8) and phosphorylated proteins (pSTAT3, pSTAT5, pAKT). The proportion of apoptotic population of bone marrow cells was determined by flow cytometry. Therefore, the data in this study will reflect the efficacy and safety of azacitidine or azacitidine combined with low-dose dasatinib in real-world maintenance therapy in patients with medium and high-risk AML.

DETAILED DESCRIPTION:
In addition to studying the overall survival, disease-free survival and recurrence rates, mortality and incidence of adverse events of patients treated with azacitidine or azacitidine combined with low-dose dasatinib, we will also study its related mechanisms. One of the pathogenesis of AML is that abnormal DNA methylation makes the cell cycle out of control and carcinogenesis by inhibiting the expression of tumor suppressor genes. In addition, the abnormal activation of tyrosine kinase signal pathway also promotes the development of leukemia. Azacitidine, the hypomethylating agents, can not only inhibit the DNA methyltransferase family, but also activate tumor suppressor genes to inhibit a variety of tyrosine kinase signaling pathways, including JAK-STAT. NaShen et al have directly demonstrated that tyrosine kinase inhibitors (TKIs) can not only inhibit the abnormal activation of tyrosine kinase pathway, but also reduce DNA methylation. This study found that the combination of the second generation TKIs and hypomethylating agents can reduce has a synergistic effect on promoting apoptosis and reducing DNA methylation. In addition, TKIs often produces drug resistance due to long exposure time, and the main mechanisms of drug resistance is due to DNA methylation and abnormal reactivation of tyrosine kinase signal pathway. The combination of TKI and azacitidine reduces DNA methylation and inhibits the reactivation of abnormal tyrosine kinase signal pathway, which is helpful to improve TKI drug resistance. Based on the above theory, we assume that patients treated with azacitidine and dasatinib may have more obvious demethylation effect, increased expression of tumor suppressive genes, more obvious apoptosis, and inhibition of phosphorylated protein expression.So we did the lab tests of these mechanisms.We innovatively used azacitidine and TKIs in the treatment of patients with AML maintenance, in order to reduce drug toxicity, enhance drug efficacy, improve patient prognosis and reduce the financial burden of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intermediate and high-risk AML who are diagnosed according to the 2016 WHO guidelines, aged ≥18 years;
2. Detect minimal residual disease(-) after induction therapy and consolidation therapy;
3. Eastern Cooperative Oncology Group (ECOG) performance status score 0-2;
4. The heart, pulmonary, liver and kidneys have sufficient organ functions:

   1. Cardiac color doppler ultrasound shows cardiac ejection fraction> 50%, heart function classification NYHA III/IV, no heart block or arrhythmia;
   2. Patients without severe restrictive/obstructive pulmonary disease;
   3. Liver function: total bilirubin (TBIL) < 2 times the upper limit of normal, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) <2.5 times the upper limit of normal;
   4. Renal function: serum creatinine (Cr) < 1.5 times the upper limit of normal.
5. The patient and family members agree and sign an informed consent form.

Exclusion Criteria:

1. Patients with malignant tumors of other organs;
2. HCV positive; or HIV positive; or one of the following HBV test results:

   1. HBsAg positive;
   2. HBsAg negative, HBcAb positive and HBV DNA titer positive;
3. Pregnant and lactating women, and patients who have family planning during the enrollment period;
4. Patients considered to be unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 30 months.
  OS is defined as the time from the date of enrollment until the date of death from any cause.
disease-free survival | up to 30 months.
  Event-free survival is defined as the time from enrollment until documented refractory disease, relapse after complete remission(CR) or CR with incomplete recovery of blood counts(CRi), or death from any cause.

SECONDARY OUTCOMES:
mortality | mortality rate at 30 months.
  The proportion of patients from enrollment to death was recorded.
recurrence rate | recurrence rate at 30 months.
  Record the proportion of patients with recurrence in the study.
adverse events | Adverse events were assessed weekly during the first and second cycles, and every two cycles thereafter (each cycle is 28 days), up to 30 months.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
apoptotic protein and phosphorylated protein | once before enrollment and once after the completion of the study, up to 30 months.
  The relative expression of apoptotic protein(caspase3, caspase8) and phosphorylated protein(pSTAT3, pSTAT5, pAKT) were detected by western blot with bone marrow aspirate.
DNA methyltransferase, tumor suppressor genes and differentiation genes | once before enrollment and once after the completion of the study, up to 30 months.
  To detect the mRNA expression of DNA methyltransferase(DNMT1, DNMT3a, DNMT3b), tumor suppressor genes(TP53,P15, P16, P21, CDH1, DOK6, SHP1, PTPN11) and differentiation gene(pu.1, C/EBPα, C/EBPβ) with bone marrow aspirate by Q-PCR.
methylation level in the promoter region of some tumor suppressor genes. | once before enrollment and once after the completion of the study, up to 30 months.
  Detection of methylation level in the promoter region of the above tumor suppressor genes by pyrophosphate sequencing using patient bone marrow aspirate.
Percentage of bone marrow cell apoptosis population | once before enrollment and once after the completion of the study, up to 30 months.
  The percentage of apoptotic population of bone marrow cells was determined by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Bei Liu, MD, Principal Investigator — The First Hospital of Lanzhou University,Lanzhou,Gansu,China
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
After the completion of the clinical trial, we will choose whether to disclose the result according to the relevant regulations of the Chinese Genetic Office.

REFERENCES:
- [Background] Tallman MS, Wang ES, Altman JK, Appelbaum FR, Bhatt VR, Bixby D, Coutre SE, De Lima M, Fathi AT, Fiorella M, Foran JM, Hall AC, Jacoby M, Lancet J, LeBlanc TW, Mannis G, Marcucci G, Martin MG, Mims A, O'Donnell MR, Olin R, Peker D, Perl A, Pollyea DA, Pratz K, Prebet T, Ravandi F, Shami PJ, Stone RM, Strickland SA, Wieduwilt M, Gregory KM; OCN; Hammond L, Ogba N. Acute Myeloid Leukemia, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jun 1;17(6):721-749. doi: 10.6004/jnccn.2019.0028. PMID 31200351
- [Background] Rashidi A, Weisdorf DJ, Bejanyan N. Treatment of relapsed/refractory acute myeloid leukaemia in adults. Br J Haematol. 2018 Apr;181(1):27-37. doi: 10.1111/bjh.15077. Epub 2018 Jan 9. PMID 29318584
- [Background] Hunault-Berger M, Maillard N, Himberlin C, Recher C, Schmidt-Tanguy A, Choufi B, Bonmati C, Carre M, Couturier MA, Daguindau E, Marolleau JP, Orsini-Piocelle F, Delaunay J, Tavernier E, Lissandre S, Ojeda-Uribe M, Sanhes L, Sutton L, Banos A, Fornecker LM, Bernard M, Bouscary D, Saad A, Puyade M, Rouille V, Luquet I, Bene MC, Hamel JF, Dreyfus F, Ifrah N, Pigneux A. Maintenance therapy with alternating azacitidine and lenalidomide in elderly fit patients with poor prognosis acute myeloid leukemia: a phase II multicentre FILO trial. Blood Cancer J. 2017 Jun 2;7(6):e568. doi: 10.1038/bcj.2017.50. No abstract available. PMID 28574488
- [Background] Tavor S, Shalit T, Chapal Ilani N, Moskovitz Y, Livnat N, Groner Y, Barr H, Minden MD, Plotnikov A, Deininger MW, Kaushansky N, Shlush LI. Dasatinib response in acute myeloid leukemia is correlated with FLT3/ITD, PTPN11 mutations and a unique gene expression signature. Haematologica. 2020 Dec 1;105(12):2795-2804. doi: 10.3324/haematol.2019.240705. PMID 33256378
- [Background] Cassileth PA, Harrington DP, Hines JD, Oken MM, Mazza JJ, McGlave P, Bennett JM, O'Connell MJ. Maintenance chemotherapy prolongs remission duration in adult acute nonlymphocytic leukemia. J Clin Oncol. 1988 Apr;6(4):583-7. doi: 10.1200/JCO.1988.6.4.583. PMID 3282032
- [Background] Molica M, Breccia M, Foa R, Jabbour E, Kadia TM. Maintenance therapy in AML: The past, the present and the future. Am J Hematol. 2019 Nov;94(11):1254-1265. doi: 10.1002/ajh.25620. Epub 2019 Sep 11. PMID 31429099
- [Background] Ades L, Itzykson R, Fenaux P. Myelodysplastic syndromes. Lancet. 2014 Jun 28;383(9936):2239-52. doi: 10.1016/S0140-6736(13)61901-7. Epub 2014 Mar 21. PMID 24656536
- [Background] Shen N, Yan F, Pang J, Zhao N, Gangat N, Wu L, Bode AM, Al-Kali A, Litzow MR, Liu S. Inactivation of Receptor Tyrosine Kinases Reverts Aberrant DNA Methylation in Acute Myeloid Leukemia. Clin Cancer Res. 2017 Oct 15;23(20):6254-6266. doi: 10.1158/1078-0432.CCR-17-0235. Epub 2017 Jul 18. PMID 28720666
- [Background] Fernandez S, Desplat V, Villacreces A, Guitart AV, Milpied N, Pigneux A, Vigon I, Pasquet JM, Dumas PY. Targeting Tyrosine Kinases in Acute Myeloid Leukemia: Why, Who and How? Int J Mol Sci. 2019 Jul 12;20(14):3429. doi: 10.3390/ijms20143429. PMID 31336846
- [Background] Amrein PC. The potential for dasatinib in treating chronic lymphocytic leukemia, acute myeloid leukemia, and myeloproliferative neoplasms. Leuk Lymphoma. 2011 May;52(5):754-63. doi: 10.3109/10428194.2011.555890. Epub 2011 Apr 4. PMID 21463117
- [Background] Gao X, Lin J, Gao L, Deng A, Lu X, Li Y, Wang L, Yu L. High expression of c-kit mRNA predicts unfavorable outcome in adult patients with t(8;21) acute myeloid leukemia. PLoS One. 2015 Apr 10;10(4):e0124241. doi: 10.1371/journal.pone.0124241. eCollection 2015. PMID 25860287
- [Background] Xie N, Zhong L, Liu L, Fang Y, Qi X, Cao J, Yang B, He Q, Ying M. Autophagy contributes to dasatinib-induced myeloid differentiation of human acute myeloid leukemia cells. Biochem Pharmacol. 2014 May 1;89(1):74-85. doi: 10.1016/j.bcp.2014.02.019. Epub 2014 Mar 4. PMID 24607273
- [Background] Al-Jamal HA, Mat Jusoh SA, Hassan R, Johan MF. Enhancing SHP-1 expression with 5-azacytidine may inhibit STAT3 activation and confer sensitivity in lestaurtinib (CEP-701)-resistant FLT3-ITD positive acute myeloid leukemia. BMC Cancer. 2015 Nov 7;15:869. doi: 10.1186/s12885-015-1695-x. PMID 26547689
- [Background] Sun GK, Tang LJ, Zhou JD, Xu ZJ, Yang L, Yuan Q, Ma JC, Liu XH, Lin J, Qian J, Yao DM. DOK6 promoter methylation serves as a potential biomarker affecting prognosis in de novo acute myeloid leukemia. Cancer Med. 2019 Oct;8(14):6393-6402. doi: 10.1002/cam4.2540. Epub 2019 Sep 4. PMID 31486300
- [Background] Lang F, Wunderle L, Pfeifer H, Schnittger S, Bug G, Ottmann OG. Dasatinib and Azacitidine Followed by Haploidentical Stem Cell Transplant for Chronic Myeloid Leukemia with Evolving Myelodysplasia: A Case Report and Review of Treatment Options. Am J Case Rep. 2017 Oct 16;18:1099-1109. doi: 10.12659/ajcr.904956. PMID 29033451
- [Background] La Rosee P, Johnson K, Corbin AS, Stoffregen EP, Moseson EM, Willis S, Mauro MM, Melo JV, Deininger MW, Druker BJ. In vitro efficacy of combined treatment depends on the underlying mechanism of resistance in imatinib-resistant Bcr-Abl-positive cell lines. Blood. 2004 Jan 1;103(1):208-15. doi: 10.1182/blood-2003-04-1074. Epub 2003 Aug 21. PMID 12933582
- [Background] Guerrouahen BS, Futami M, Vaklavas C, Kanerva J, Whichard ZL, Nwawka K, Blanchard EG, Lee FY, Robinson LJ, Arceci R, Kornblau SM, Wieder E, Cayre YE, Corey SJ. Dasatinib inhibits the growth of molecularly heterogeneous myeloid leukemias. Clin Cancer Res. 2010 Feb 15;16(4):1149-58. doi: 10.1158/1078-0432.CCR-09-2416. Epub 2010 Feb 9. PMID 20145167
- [Background] Patel AB, Pomicter AD, Yan D, Eiring AM, Antelope O, Schumacher JA, Kelley TW, Tantravahi SK, Kovacsovics TJ, Shami PJ, O'Hare T, Deininger MW. Dasatinib overcomes stroma-based resistance to the FLT3 inhibitor quizartinib using multiple mechanisms. Leukemia. 2020 Nov;34(11):2981-2991. doi: 10.1038/s41375-020-0858-1. Epub 2020 May 14. PMID 32409689